CLINICAL TRIAL: NCT03532165
Title: Use of Bedside Ultrasound in Emergency Department Patients With Concern for Pulmonary Embolism to Reduce CT Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Dorcas Boahema Pinto, Dr., Albany Medical College
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 4975
Record Dates: First submitted 2018-05-01; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis Leg; Ultrasound Imaging
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: In all enrolled patients with concern for pulmonary embolism, a lower extremity ultrasound will be performed at the patient's bedside by the emergency room provider. If it is positive for a deep vein thrombosis, then a confimatory ultrasound will be performed by the vascular lab, and the patient started on anticoagulation to treat both the DVT and presumed PE. No CTA will be obtained in this group. Everyone else who had a negative bedside ultrasound performed by the ER provider will not receive a second ultrasound, but will rather go on to get the CT angiogram of the chest they would have likely received if not in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive lower extremity ultrasound (Other): This group found to to have a deep venous thrombosis on lower extremity ultrasound will not have a CT of the chest ordered from the emergency department, and will be treated for the DVT and presumed PE.
  Interventions: Diagnostic Test: Lower extremity Ultrasound
- Negative lower extremity ultrasound (Other): This group that does not have a deep venous thrombosis on lower extremity ultrasound will proceed to get the CT of the chest .
  Interventions: Diagnostic Test: Lower extremity Ultrasound

INTERVENTIONS:
Diagnostic Test: Lower extremity Ultrasound — One group may forego a CT angiogram of the chest if they have a positive lower extremity ultrasound. The other group with a negative ultrasound may still require CT angiogram imaging.
  Other Names: CT angiogram of the chest

SUMMARY:
At most institutions, the average patient with clinical concern for PE(pulmonary embolism) will have a CT angiogram(CTA) with contrast of the lungs performed to evaluate for a clot. However, CTA has risks including contrast- induced allergic reactions and nephropathy, as well as radiation which has been linked to development of cancer later in life. There is literature that has looked at using lower extremity doppler ultrasound first to evaluate for a DVT (deep venous thrombosis) in patients where there is concern for a PE. There is also literature showing that emergency medicine physicians can perform adequate lower extremity compression ultrasounds (LCUS), at the bedside with results similar to that of the ultrasound tech. The goal of this project is to fuse both principles by having emergency medicine physicians perform LCUS at the bedside, to help reduce CTA utilization in the evaluation of PE.

DETAILED DESCRIPTION:
In this study, the subgroup of hemodynamically stable patients felt to be at moderate to high risk for PE will receive a bilateral LCUS before possible CTA/VQ imaging. The LCUS of the entire proximal leg including the popliteal fossa will be performed by an emergency medicine resident provider in conjunction with their attending. All positive studies will then be confirmed with a second ultrasound by the Albany Medical Center's vascular laboratory service. Patients with confirmed acute positive studies identifying a DVT will be treated for a presumed PE, which is the same treatment as that for the DVT. No CTA will be ordered from the ED. They will be anticoagulated and admitted to the hospital, with further management as per the inpatient hospital team. Patients with a negative emergency department LCUS done by the resident will receive either a CTA or a VQ (ventilation/perfusion) scan as per the initial treatment plan established by the attending physician.

According to this protocol, patients discharged home by default must have had a negative CTA or VQ scan, and so PE was effectively ruled out. Therefore they will not require further follow up after discharge. However, we will follow patients who were admitted throughout their admission course. Through review of medical records, we will take note of any complications such as any issues with starting anticoagulation treatment without a CTA, misdiagnoses, whether a CTA was ordered later as a part of their course and why, and further details.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Concern for PE (moderate to high risk) that warrants imaging of the chest

Exclusion Criteria:

* Age less than 18
* nidus for DVT in upper extremity (eg. PICC (peripherally inserted central Cather) line, etc)
* already anti-coagulated at presentation
* above the knee- leg cast
* prisoners
* DVT ultrasound or CTA prior to presentation
* Hemodynamically unstable:
* SBP (systolic blood pressure) <90 for >15min
* Drop of SBP by at least 40mmHG for >15mins
* Organ hypoperfusion (eg cold extremities, mental confusion, low urine outpt <30cc/hr, etc
* need for pressors
* Other concerns in thorax necessitating inevitable CT chest imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-02-22 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Absolute reduction in CT imaging to diagnose PE | for duration of the study,about 1 year
  With the use of lower extremity ultrasound to diagnose DVT, some patients may forego the need for CT imaging while receiving appropriate care/treatment.

SECONDARY OUTCOMES:
Potential reduction in CT imaging to diagnose PE | for duration of the study, about 1 year
  If a CT is ordered on a patient with a positive lower extremity ultrasound by an inpatient physician later during the admission, we will calculate what the reduction in CT imaging would have been if the protocol had been followed to the end.
Time to start of treatment | for duration of the study , about 1 year
  The use of bedside ultrasound may allow for making a diagnoses more quickly, and therefore potentially starting treatment sooner.
Cost-analysis | for duration of study, about 1 year
  The use of ultrasound may have less cost than using a CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Dorcas B Pinto, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center Department of Emergency Medicine, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skinner S. Pulmonary embolism: assessment and imaging. Aust Fam Physician. 2013 Sep;42(9):628-32. PMID 24024223
- [Background] Da Costa Rodrigues J, Alzuphar S, Combescure C, Le Gal G, Perrier A. Diagnostic characteristics of lower limb venous compression ultrasonography in suspected pulmonary embolism: a meta-analysis. J Thromb Haemost. 2016 Sep;14(9):1765-72. doi: 10.1111/jth.13407. Epub 2016 Aug 17. PMID 27377039
- [Background] Perrier A, Roy PM, Aujesky D, Chagnon I, Howarth N, Gourdier AL, Leftheriotis G, Barghouth G, Cornuz J, Hayoz D, Bounameaux H. Diagnosing pulmonary embolism in outpatients with clinical assessment, D-dimer measurement, venous ultrasound, and helical computed tomography: a multicenter management study. Am J Med. 2004 Mar 1;116(5):291-9. doi: 10.1016/j.amjmed.2003.09.041. PMID 14984813
- [Background] Poley RA, Newbigging JL, Sivilotti ML. Estimated effect of an integrated approach to suspected deep venous thrombosis using limited-compression ultrasound. Acad Emerg Med. 2014 Sep;21(9):971-80. doi: 10.1111/acem.12459. PMID 25269577